CLINICAL TRIAL: NCT06217822
Title: A Phase 1 Open-label, First-in-human, Multi-center Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of 225Ac-PSMA-Trillium in Participants With Advanced Metastatic Castration-resistant Prostate Cancer (mCRPC)
Brief Title: First-in-human Study of 225Ac-PSMA-Trillium (BAY 3563254) in Participants With Advanced Metastatic Castration-resistant Prostate Cancer (mCRPC)
Acronym: PAnTHA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22049; 2023-507486-26-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-12-19; First posted 2024-01-23 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Advanced Metastatic Castration-resistant Prostate Cancer; Prostate Specific Membrane Antigen (PSMA) Expression
Keywords: mCRPC; PSMA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Dose escalation of BAY3563254 (Experimental): Participants with advanced mCRPC will receive increased 225Ac-PSMA-Trillium doses in a planned stepwise fashion.
  Interventions: Drug: 225Ac-PSMA-Trillium (BAY3563254)
- Dose expansion group A of BAY3563254 (Experimental): Participants with advanced mCRPC must have received at least 1 but no more than 2 prior taxane-based chemotherapy regimens. No prior treatment with 177Lu-PSMA.
  Interventions: Drug: 225Ac-PSMA-Trillium (BAY3563254)
- Dose expansion group B of BAY3563254 (Experimental): Participants with advanced mCRPC must *not* have received taxane-based chemotherapy since becoming castration resistant. No prior treatment with 177Lu-PSMA.
  Interventions: Drug: 225Ac-PSMA-Trillium (BAY3563254)
- Dose expansion group C of BAY3563254 (Experimental): Participants with advanced mCRPC treated with 225Ac-PSMA-Trillium, who have received treatment with an established 177Lu-PSMA therapy and who did not discontinue 177Lu-PSMA treatment due to intolerance.
  Interventions: Drug: 225Ac-PSMA-Trillium (BAY3563254)
- 225Ac-PSMA-Trillium Imaging and Dosimetry (Experimental): The 225Ac-PSMA-Trillium Imaging and Dosimetry Substudy will enroll throughout both dose escalation and dose expansion, starting with the first dose level in dose escalation. The substudy will generally be available at all study sites to participants in the main study.
  Interventions: Drug: 225Ac-PSMA-Trillium (BAY3563254)
- HPGe or NaI Whole Body Radioactivity Measurement of 225Ac-PSMA-Trillium (Experimental): HPGe or NaI measurements of whole-body radioactivity of 225Ac and its daughters as a function of time will be conducted on an optional basis during dose escalation and dose expansion at selected sites to evaluate the clearance of total radioactivity from the body over time. Participants in the 111In-PSMA-Trillium and Tris-POC Imaging Substudy will not be eligible for this HPGe or NaI Whole Body Radioactivity Measurement of 225Ac-PSMA-Trillium Substudy.
  Interventions: Drug: 225Ac-PSMA-Trillium (BAY3563254)

INTERVENTIONS:
Drug: 225Ac-PSMA-Trillium (BAY3563254) — Intravenous slow injection on Day 1 of a 6 week treatment cycle.

SUMMARY:
Researchers are looking for a better way to treat participants who have metastatic castration-resistant prostate cancer (mCRPC).

mCRPC is a cancer of the prostate (male reproductive gland found below the bladder) that has spread to other parts of the body. This type of prostate cancer does not respond to hormone treatment used to lower the level of testosterone, a male sex hormone, to prevent cancer from growing.

The study treatment 225Ac-PSMA-Trillium, also called BAY3563254, is under development to treat advanced metastatic castration-resistant prostate cancer. It works by binding to PSMA and giving off radiation that can damage cancer cells and stop them from growing.

The main purpose of this first-in-human study is to learn:

* How safe is BAY3563254 in participants.
* What is the recommended dose of BAY3563254 that is safe and works well that will be further tested in Part 2 of the study.
* How well does BAY3563254 work in participants.

To answer this, the researchers will look at:

* The number and severity of medical problems including serious medical problems that participants experience after taking BAY3563254
* The number of dose-limiting toxicities (DLT) at each dose level. A DLT is a medical problem caused by a drug that is too severe to continue the use of that specific dose.
* The number of participants whose cancer completely disappears (complete response) or reduces by at least 30% (partial response) after taking the treatment (also known as objective response rate (ORR))
* The number of participants who have a decrease in the levels of PSA* by at least 50% in their blood (also known as PSA50). PSA is a protein made by the prostate gland. High levels of PSA may indicate the presence of prostate cancer.
* Participants' best response to treatment based on their PSA levels (also known as the best overall PSA response).

The study will have two parts. The first part, called dose escalation, is done to find the most appropriate dose of BAY3563254 for use in the second part of the study. For this, each participant will receive one of different increasing amounts of BAY3563254. They will take BAY3563254 as an injection into a vein. All participants in the second part of the study, called dose expansion, will receive the most appropriate dose of BAY3563254 that was identified from the first part of the study.

Participants in this study will take the study treatment once every 6 weeks, which is known as a treatment cycle. Each participant will have up to 4 of these treatment cycles, if the participant benefits from the treatment. Each participant will be in the study for approximately 6 years, including a screening phase of up to 30 days, 6 months of treatment depending on the participant's benefit, and a follow up phase of 60 months after the end of treatment.

In addition, substudies performed during both dose escalation and dose expansion parts of the study will evaluate:

* the clearance of radioactivity from the body over time
* the doses of radiation that are delivered to normal organs and tumors

During the study, the doctors and their study team will:

* take blood and urine samples
* check vital signs such as blood pressure, heart rate, and body temperature
* examine heart health using electrocardiogram (ECG)
* take tumor samples if required
* check if the participants' cancer has grown and/or spread using CT (computed tomography) or MRI (magnetic resonance imaging) and bone scan
* check the tumor status using PET (positron emission tomography)
* check the amount of radiation absorbed by tumors and normal organs using SPECT/CT (single-photon emission tomography and computed tomography scan)
* ask the participants questions about how they are feeling and what adverse events they are having.

An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events, irrespective if they think it is related or not to the study treatments. In addition, the participants will be asked to complete a questionnaire on quality of life at certain time points during the study.

The treatment period ends with a visit in 6-12 weeks after the last BAY3563254 dose. About 6-12 weeks after the last dose and every 6 weeks thereafter, the study doctors and their team will check the participants' health and any changes in their cancer. This active follow-up period ends after 18 months. The long-term follow-up period will start after the end of the active follow-up visit and will continue for up to 60 months after the the last BAY3563254 dose. Participants will be contacted, typically by phone call or clinic visit, approximately every 12 weeks after the end of active follow-up.

ELIGIBILITY:
Inclusion Criteria:

* mCRPC with pathological confirmation of adenocarcinoma without small-cell or neuroendocrine features.
* Previous treatment with at least 1 novel androgen axis drug (NAAD) (e.g., enzalutamide, apalutamide, darolutamide and/or abiraterone).
* Prior orchiectomy and/or ongoing androgen deprivation therapy and a castrate level of serum testosterone (<50 ng/dL or <1.7 nmol/L).
* Prior taxane treatment:

  * Dose Escalation: Participants must either have had prior treatment with at least 1 but no more than 2 taxane regimens, or been deemed ineligible for or refused taxane therapy on consultation with their physician
  * Dose Expansion Group A: Participants must have had prior treatment with at least 1 but no more than 2 taxane regimens, in the castration-resistant setting
* Dose Expansion Group B: Participants must not have received any taxane regimens since becoming castration-resistant

  * Dose Expansion Group C: Participants must either have had prior treatment with at least 1 but no more than 2 taxane regimens, or been deemed ineligible for or refused taxane therapy on consultation with their physician
* Prior treatment with an established Lu-PSMA therapy (i.e., dose activity and cycles comparable to approved treatments) is required for participants in Dose Expansion Group C only. More specifically, to qualify for this expansion group, participants must not have discontinued 177Lu-PSMA treatment due to intolerance.
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1.
* Adequate bone marrow, hepatic, and renal function, as assessed by the following laboratory requirements within 30 days before start of study intervention, as indicated below. Note that blood transfusions (red blood cells or platelets) and administration of G-CSF or GM-CSF are prohibited within 21 days prior to screening for the below bone marrow-related parameters.

  * Hemoglobin ≥9.0 g/dL
  * Absolute neutrophil count (ANC) ≥1500/mm^3
  * Platelet count ≥100,000/mm^3
  * Total bilirubin ≤1.5 x the Upper limit of normal (ULN), or ≤3×ULN if the participant has a confirmed history of Gilbert's syndrome (note that participants with Gilbert's syndrome should be carefully evaluated for other liver-related disorders that may impact their suitability for this study).
  * Alanine transaminase (ALT) and Aspartate transaminase (AST) ˂2.5 x ULN (≤5 x ULN for participants with liver involvement)
  * Participants on a stable dose of anticoagulation therapy are allowed to participate if they have no sign of bleeding or clotting, and prothrombin time international normalized ratio (PT/INR) and activated partial thromboplastin time (aPTT) test results are acceptable at the Investigator's discretion
  * Estimated glomerular filtration rate (eGFR) >60 mL/min/1.73 m^2, according to the Modified Diet in Renal Disease (MDRD) abbreviated formula and serum creatinine ≤1.5 x ULN
* Participants must have at least one PSMA-positive (prostate-specific membrane antigen) distant metastatic lesion on the screening PSMA PET/CT scan using the study-designated PSMA PET tracers, as determined by the site Investigator. For eligibility purposes, a PSMA-positive lesion must have activity greater than the liver by visual assessment of the screening PSMA PET/CT. A PSMA-positive metastatic lesion should not correspond to a normal tissue structure or benign lesion.
* Documented progressive mCRPC per PCWG3, and a minimum starting PSA value of 2.0 ng/mL is mandatory. Progressive mCRPC is defined as meeting at least one of the following criteria:

  1. PSA progression (defined as 2 consecutive increases over a previous reference value obtained at a minimum of 1-week
  2. Radiological progression in soft-tissue lesions according to PCWG3 modification of RECIST v1.1 criteria
  3. Progression of bone disease (defined as ≥ 2 new bone lesions according to PCWG3 bone scan criteria)

Exclusion Criteria:

* Participants who have any of the following tumor lesions which are PSMA negative AND meet the size criteria below are excluded as determined by the site Investigator. A PSMA-negative lesion for eligibility purposes must have activity equal to or less than the liver by visual assessment of the screening PSMA PET/CT scan using the study-designated PSMA PET/CT tracers. A PSMA-negative metastatic lesion should not correspond to a normal tissue structure or benign lesion.

  * a. Any single or multiple lymph node(s) ≥2.5 cm in the short axis.
  * b. Any solid organ metastasis (e.g., lung, liver, adrenal glands, etc.) that is ≥1 cm in the short axis.
  * c. Any bone metastasis with a soft tissue component ≥ 1 cm in short axis with the soft tissue component being PSMA-negative. PSMA-negative osseous metastases without a soft tissue component do not exclude a participant.
  * d. Predominantly necrotic lesions with greater than 1 cm of enhancing tissue on contrast-enhanced computed tomography / magnetic resonance imaging (CT/MRI).
* Prior systemic anticancer therapy including chemotherapy, NAAD, biologic therapy, immunotherapy, or investigational therapies within 4 weeks of the start of study treatment, except luteinizing hormone-releasing hormone (LHRH) or gonadotropin-releasing hormone (GnRH). Start of study treatment is allowed in shorter timeframes if 5 half-lives of the prior drug(s) have elapsed.
* Prior radiopharmaceutical treatment using actinium-225.

Other prior radiopharmaceutical treatments:

* Dose escalation and Dose expansion Groups A and B: Prior treatment with a radiopharmaceutical is prohibited, with the exception of prior treatment with radium-223 dichloride more than 3 months before the start of study intervention. Note: Participants who have discontinued radium-223 dichloride treatment due to intolerance are excluded from Groups A and B.
* Dose expansion Group C: Prior treatment with a radiopharmaceutical is prohibited with the following exceptions: Prior treatment with radium-223 dichloride more than 3 months before the start of study intervention is permitted; and prior treatment with 177Lu-PSMA more than 6 weeks before the start of study intervention is required. Note: Participants who have discontinued 177Lu-PSMA or radium-223 dichloride treatment due to intolerance are excluded from Group C.

  * Prior definitive therapy (radiotherapy or surgery) completed less than 6 weeks before the start of study intervention. Note that palliative radiotherapy completed less than 6 weeks before the start of study intervention will be allowed if: (i) no more than 10% of the participants' bone marrow is irradiated, (ii) it does not encompass all potential target/measurable lesions for participants in dose expansion.
  * Toxic effects of Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Grade ≥2 from prior anticancer therapy not yet stabilized or where significant post-treatment toxicities have been observed. Chronic toxic effects of CTCAE Grade ≤2 from prior anticancer therapy where no further resolution is expected do not require exclusion with agreement between the Investigator and Sponsor (e.g., chemotherapy-induced neuropathy, fatigue, alopecia, anorexia, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2027-06-14 (Estimated); Study Completion 2031-05-24 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation and Dose Expansion: Incidence of TEAEs (including TESAEs) | After the first administration of study intervention up to 42 days after the last dose of study intervention
  TEAE: Treatment-emergent adverse event TESAE: Treatment-emergent serious adverse event
Dose Escalation and Dose Expansion: Severity of TEAEs (including TESAEs) | After the first administration of study intervention up to 42 days after the last dose of study intervention
Dose Escalation: Incidence of DLTs | Up to and including Cycle 3 (each cycle is 42 days)
  DLT: Dose-Limiting Toxicities
Dose Escalation and Dose Expansion: ORR by PCWG3 guideline based on Investigator review | Up to 18 months after end of treatment
  ORR is defined as the proportion of participants who have a confirmed complete response (CR) or partial response (PR) per PCWG3 guidelines as assessed by the Investigator.
Dose Escalation and Dose Expansion: PSA50 response | At 12 weeks or later (up to 18 months after end of treatment)
  PSA50 response is defined as a ≥50% decline in PSA value from baseline (Cycle 1 Day 1).
Dose Expansion: Best overall PSA response | Up to 18 months after end of treatment
  Best overall PSA response corresponds to the maximum percentage decline or the minimum percentage increase (if no decline) in PSA value from baseline (Cycle 1 Day 1).

SECONDARY OUTCOMES:
Dose Expansion: Recommended dose for further clinical development | Up to 18 months after end of treatment
Dose Expansion: Recommended dose regimen for further clinical development | Up to 18 months after end of treatment
Dose Escalation and Dose Expansion: Radiologic progression-free survival (rPFS) by PCWG3 based on Investigator review | Up to 18 months after end of treatment
  rPFS is defined as the time from the start of study treatment to the date of first observed disease progression (Investigator's radiological assessment by PCWG3) or death due to any cause, if death occurs without progression is documented.
Dose Escalation and Dose Expansion: Duration of response (DOR) by PCWG3 based on Investigator review | Up to 18 months after end of treatment
  DOR is defined as the time from the first documented objective response of PR or CR by PCWG3, whichever occurs earlier, to disease progression or death (if death occurs without progression is documented).
Dose Escalation and Dose Expansion: Duration of PSA50 response | Up to 18 months after end of treatment
  Duration of PSA50 response is defined as the time from the first documented PSA50 response to PSA progression by PCWG3 or death (if death occurs without progression is documented).
Dose Escalation and Dose Expansion: Cmax of 225Ac | Cycle 1, cycle 2 (From pre-dose up to Day 36 post-dose for each cycle)
Dose Escalation and Dose Expansion: AUC and AUC(0-tlast) of 225Ac | Cycle 1, cycle 2 (From pre-dose up to Day 36 post-dose for each cycle)
Dose Escalation and Dose Expansion: Cmax of PSMA-Trillium-macropa peptide | Cycle 1, cycle 2 (From pre-dose up to Day 36 post-dose for each cycle)
Dose Escalation and Dose Expansion: AUC and AUC(0-tlast) of PSMA-Trillium-macropa peptide | Cycle 1, cycle 2 (From pre-dose up to Day 36 post-dose for each cycle)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (4):
  - City of Hope - Duarte Cancer Center, Duarte, California
  - M Health Fairview Masonic Cancer Clinic - Clinics and Surgery Center, Minneapolis, Minnesota
  - XCancer Omaha, Omaha, Nebraska
  - The University of Texas MD Anderson Cancer Center - Texas Medical Center, Houston, Texas
- Belgium (3):
  - Institut Jules Bordet / Nuclear Medicine, Anderlecht
  - AZ Groeninge Campus Kennedylaan - Urology, Kortrijk
  - UZ Leuven - Campus Gasthuisberg - Nuclear Medicine, Leuven
- Canada (7):
  - Cross Cancer Institute, Clinical Trials Unit, Edmonton, Alberta
  - BC Cancer - Vancouver Site, Vancouver, British Columbia
  - Juravinski Cancer Centre - Clinical Trials Department, Hamilton, Ontario
  - Princess Margaret Cancer Centre - University Health Network - Department of Medical Oncology and Hematology, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - McGill University Health Centre (MUHC) - Research Institute (RI) - McConnell Centre for Innovative Medicine (CIM), Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke (CHUS) - Hopital Fleurimont, Sherbrooke, Quebec
- Finland (5):
  - Kuopio University Hospital, Kuopion yliopistollinen sairaala (KYS) - Syövänhoitokeskus, Kuopio, Northern Savonia
  - HUS-Yhtymä, Helsingin yliopistollinen sairaala (HUS) - Syöpäkeskus, Helsinki, Uusimaa
  - Docrates Mehiläinen Syöpäsairaala, Helsinki, Uusimaa
  - Tampere University Hospital, Tampereen yliopistollinen sairaala (TAYS) - Syöpäkeskus, Tampere
  - Turku University Hospital, Turun yliopistollinen sairaala (TYKS), Turku
- Italy (2):
  - Istituto Europeo di Oncologia s.r.l - Medicina Nucleare, Milan
  - IRCCS Istituto Nazionale Tumori Fondazione Pascale - S. C. Medicina Nucleare e Terapia Metabolica, Napoli
- Netherlands (2):
  - Universitair Medisch Centrum Groningen (UMCG) - UMC Groningen Comprehensive Cancer Center, Groningen
  - Erasmus Medisch Centrum, Rotterdam
- Sweden (4):
  - Sahlgrenska Universitetssjukhuset - Klinisk prövningsenhet Fas I/FIH, Gothenburg
  - Skånes Universitetssjukhus Lund - Onkologens kliniska forskningsenhet, Lund
  - Karolinska Universitetssjukhuset - Fas I-enheten Solna CKC, Stockholm
  - Akademiska Sjukhuset - Fas-I-enheten, Uppsala
- Switzerland (3):
  - Kantonsspital Baden, Baden, Canton of Aargau
  - Universitätsspital Basel, Basel, Canton of Basel-City
  - Univestitätsspital Zürich (USZ), Zurich
- United Kingdom (3):
  - University College London Hospitals NHS Foundation Trust | University College Hospital - NIHR UCLH Clinical Research Facility, London, Greater London
  - The Royal Marsden NHS Foundation Trust | Sutton - Oak Foundation Drug Development Unit, Sutton, Surrey
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust | Freeman Hospital - Cancer Trials Research Centre, Newcastle upon Tyne, Tyne and Wear

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.